CLINICAL TRIAL: NCT03000764
Title: Study of RNA and Heat Shock Protein (HSP) Derived Biomarkers in Radiation-induced Fibrosis in Patients Treated for Breast Cancer.
Brief Title: RNA and Heat Shock Protein Biomarkers in Radiation-induced Fibrosis in Breast Cancer
Acronym: SPLICI-Rad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A00592-49
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Carcinoma; Fibrosis
Keywords: Skin biopsy; Radiotherapy; RNA biomarker; HSP biomarker; Exon junction array; Gene expression; Radiosensitivity prediction
MeSH Terms: conditions — Breast Neoplasms; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarkers (Experimental)
  Interventions: Other: skin biopsies; Other: blood samples

INTERVENTIONS:
Other: skin biopsies — Biopsies (12 G) will be performed :
  * in non-irradiated breast skin
  * in irradiated breast skin
Other: blood samples — blood samples are collected:
  * 10 ml in EDTA tube
  * 2,5 ml in PAXgene Blood RNA tube
  * 4 ml in EDTA tube

SUMMARY:
The purpose of this study is to seeking a molecular signature of pathological radiation induced fibrosis based on the response of skin fibroblasts after irradiation, comparing two groups of patients distinguished by their individual radiosensitivity. The signature will integrate recent insights in terms of alternative splicing of mRNAs and level of expression of non-coding RNAs, particularly long non-coding RNAs, snRNAs, snoRNAs and microRNAs. In each group each expression patterns of candidate HSP proteins potentially predictive of pathological radiation induced fibrosis (HSP27, HSP70, αβ crystalline) in the serum and on cell culture will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* women
* age ≥ 18 and <70 years old
* non metastatic disease
* ECOG performance status 0 or 1
* chest size ≤ 110 cm et bra size <D
* absence of reconstructive breast surgery
* patient able to undergo blood samples (haematological conditions allowing blood sample)
* non-evolving carcinological disease
* absence of systemic inflammatory disease (other than scleroderma) or diabetes
* no inflammatory ou infectious flare on biopsy site at the time of inclusion
* invasive or in situ breast carcinoma
* ability to provide an informed written consent form
* affiliation to a social security system

Then stratification into two groups :

group 1 : radio-sensitive patients

* Post-operative radiotherapy completed at least 6 months ago AND
* radiation induced dermal and/or soft tissue toxicity (dermatitis, fibrosis, atrophy) rated > 2 (CTCAE v4.0 scale)

group 2 : radio-tolerant (control) patients

* Post-operative radiotherapy completed more than 4 years ago AND
* radiation induced dermal and/or soft tissue toxicity (dermatitis, fibrosis, atrophy) rated ≤1 (CTCAE v4.0 scale) .

Exclusion Criteria:

* age <18 or > 70 years old
* evolutive cancer / metastatic disease
* chest size > 110 cm et bra size ≥ D
* previous reconstructive breast surgery
* ECOG performance status > 1
* systemic inflammatory disease or diabetes
* inflammatory ou infectious flare on biopsy site at the time of inclusion, very significant ulceration in the treated breast
* anemic patients
* use of oral anticoagulants
* pregnant or likely to be in 6 months
* patients deprived of liberty or under supervision
* non-affiliation to a social security system

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Global mRNA alternative splicing and expression of non-coding RNAs profiles in healthy dermal fibroblasts | 6 months
  frequency of inclusion of individual exons within the set of mRNA isoforms (overall splicing profile) and variation in expression of non-coding RNAs

SECONDARY OUTCOMES:
Transcriptomic signature of pathological induced fibrosis when comparing the primary outcome between the two populations on cultured fibroblasts | 6 months
Transcriptomic signature of pathological induced fibrosis when comparing the primary outcome between the two populations on serum | 6 months
Individual radiosensitivity on healthy dermal fibroblasts | 6 months
  The micronuclei will be counted 24 hours after ex vivo irradiation with an indirect immunofluorescence assay (53BP1 + pATM antibodies)
Comparison of the overall mRNA splicing and non-coding RNA expression profiles between non irradiated and irradiated dermal fibroblasts in the same individual | 6 months
Changes in cellular distribution of the main non-coding RNAs whose expression varies significantly within the pre-identified signature between the 2 groups of patients | 6 months
  The cellular distribution is defined as the compartment (nucleoplasm, nucleolus, intra-nuclear corpuscles, cytosol, RE, mitochondria ...) marked by the fluorescent probe labeled to the non-coding RNAs of interest (RNA-FISH)
seric HSP proteins potentially predictive of pathological induced fibrosis | 6 months
  HSP27, HSP70 and αB crystalline measured in serum with ELISA assay
Cellular distribution of specific HSP on fibroblast culture in each group of patients | 6 months
  immunolabeling of HSPs and spatial mapping and sub-nuclear distributions
Potential interactions between DNA damage response proteins and candidate HSP | 6 months
  Collocation of HSPs with pATM and 53-BP1 (confocal microscopy / FLIM)

CONTACTS AND LOCATIONS:
Overall Officials: VOGIN GUILLAUME, MD, PhD, Principal Investigator — Institut de Cancérologie de Lorraine; BEHM-ANSMANT Isabelle, PhD, Principal Investigator — UMR 7365 CNRS-Université de Lorraine, IMoPA
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No